CLINICAL TRIAL: NCT02261272
Title: Internet-based Treatment for Insomnia in Norway.
Brief Title: Internet-based Treatment for Insomnia
Acronym: SHUTiNorse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Borge Sivertsen, Professor, Norwegian Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHUTiNorse
Record Dates: First submitted 2013-11-01; First posted 2014-10-10 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Psychophysiologic Insomnia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CBT for insomnia (Experimental): Cognitive-behavioral therapy for insomnia
  Interventions: Behavioral: CBT for insomnia SHUTi
- Sleep Hygiene (Active Comparator): Psychoeducational intervention based on standard sleep hygiene advices
  Interventions: Behavioral: passive patient education/sleep hygiene

INTERVENTIONS:
Behavioral: CBT for insomnia SHUTi — SHUTi
  Arms: CBT for insomnia
Behavioral: passive patient education/sleep hygiene
  Arms: Sleep Hygiene

SUMMARY:
The study will test an internet-based treatment for insomnia.

DETAILED DESCRIPTION:
This study will develop and evaluate the feasibility of a cost-effective, more accessible alternative treatment approach for insomnia. Traditional CBT, including the behavioral, cognitive, and educational aspects, will be operationalized and transformed for an Internet intervention system, so individuals can access a personalized treatment any time, at their own convenience. Phase 1 of this study will involve developing the web program. The investigators research team and collaborators has extensive experience developing such web interventions, as well as considerable experience with insomnia. Phase 2 will be a large randomized controlled trial testing the Internet intervention compared to passive patient education/sleep hygiene. Two hundred individuals with insomnia will be assessed pre and post the six week treatment program. It is hypothesized that the Internet intervention will promote improvements in sleep, mood, and cognitive functioning. If successful, the current project may result in improved implementation of a low-threshold treatment for a common disorder with devastating impact on both individual and socioeconomic outcomes

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. fulfillment of the DMS-IV criteria for insomnia
3. duration of at least 3 months
4. complaints of impaired daytime functioning

Exclusion Criteria:

1. presence of a major depressive disorder or other severe mental disorder as identified by in the telephone interview
2. working night shifts and unable to discontinue this work pattern
3. having a serious somatic condition preventing further participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Insomnia symptoms | Assessment points: pre- and post-treatment (6 weeks after baseline), and 6 and 18 month FU
  Self-reported questionnaires (Berge Insomnia Scale and Insomnia Severity Index)): change from baseline to post-treatment and FU

SECONDARY OUTCOMES:
Daytime functioning (mental health problems and fatigue) | Assessment points: pre- and post-treatment (6 weeks after baseline), and 6 and 18 month FU
  Self-reported questionnaires
Sleep diary data | Assessment points: pre- and post-treatment (6 weeks after baseline), and 6 and 18 month FU
  Sleep duration, sleep onset latency and nocturnal wake time: change from baseline to post-treatment and FU

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Institute of Public Health, Bergen, Norway

REFERENCES:
- [Derived] Lien M, Bredeli E, Sivertsen B, Kallestad H, Pallesen S, Smith ORF, Faaland P, Ritterband LM, Thorndike FP, Vedaa O. Short and long-term effects of unguided internet-based cognitive behavioral therapy for chronic insomnia in morning and evening persons: a post-hoc analysis. Chronobiol Int. 2019 Oct;36(10):1384-1398. doi: 10.1080/07420528.2019.1647435. Epub 2019 Aug 1. PMID 31368382
- [Derived] Vedaa O, Hagatun S, Kallestad H, Pallesen S, Smith ORF, Thorndike FP, Ritterband LM, Sivertsen B. Long-Term Effects of an Unguided Online Cognitive Behavioral Therapy for Chronic Insomnia. J Clin Sleep Med. 2019 Jan 15;15(1):101-110. doi: 10.5664/jcsm.7580. PMID 30621837
- [Derived] Hagatun S, Vedaa O, Harvey AG, Nordgreen T, Smith ORF, Pallesen S, Havik OE, Thorndike FP, Ritterband LM, Sivertsen B. Internet-delivered cognitive-behavioral therapy for insomnia and comorbid symptoms. Internet Interv. 2018 Feb 21;12:11-15. doi: 10.1016/j.invent.2018.02.003. eCollection 2018 Jun. PMID 30135764